CLINICAL TRIAL: NCT03532867
Title: Study of Changes in Retrofoveolar Choroidal Thickness Measured by Optical Coherence Tomography During Aerobic Exercise Inducing an Increase in Systolic Blood Pressure in Healthy Subjects
Brief Title: Study of Changes in Retrofoveolar Choroidal Thickness During Aerobic Exercise
Acronym: MOPAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0059; 2017-A02206-47 (Other: ID-RCB)
Record Dates: First submitted 2018-04-16; First posted 2018-05-22 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Choroid Disease; Hypertension Ocular
Keywords: Exercise Test; Blood Pressure; Choroid
MeSH Terms: conditions — Choroid Diseases; Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: To study the changes in choroidal thickness of the macular region during aerobic exercise inducing an increase in systolic and diastolic blood pressure in healthy subjects measured by Optical Coherence Tomography (OCT) provides cross-sectional imaging of the choroid and in vivo measurement of its thickness Patients are treated in the usual way but the study is an interventional study, with minimal risks and constraints, because of the imaging (OCT image in EDI mode)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): After an ophthalmic consultation, the healthy volunteers are summoned to perform the exercise test in the form of an aerobic exercise on an ergometric bicycle with 3 different intensity levels calculated on the theoretical maximum aerobic power.
  The OCT examination in the EDI mode, centered on the macular and peri-papillary region, as well as the systolic and diastolic blood pressure and the heart rate.
  In healthy patients performing aerobic physical exercise in the Department of Sports Medicine , the investigators will perform the following Intervention :
  * Examination of pressures before stopping the exercise
  * Examination of pressure during the exercise
  * Examination of pressures after stopping the exercise
  Interventions: Other: Examination of pressures before stopping the exercise; Other: Examination of pressure during the exercise; Other: Examination of pressures after stopping the exercise

INTERVENTIONS:
Other: Examination of pressures before stopping the exercise — In healthy volunteers performing aerobic physical exercise in the Department of Sports Medicine, the investigators will perform different examinations :
  * Macular and peri-papillary OCT in EDI mode (bilateral examination),
  * Intraocular pressure (bilateral examination)
  * Measurement of systolic and diastolic blood pressure
  * Heart rate measurement Exercise testing will be performed on bicycle measuring session with 10 minutes at moderate intensity ( 30% OF MPA), 10 minutes at sustained intensity ( 50% of MPA) and 3 minutes at maximum (70% of MPA).
  The theoretical maximal aerobic power was calculated by a mathematical formula.
Other: Examination of pressure during the exercise — In healthy volunteers performing aerobic physical exercise in the Department of Sports Medicine, the investigators will perform different examinations :
  * Macular and peri-papillary OCT in EDI mode (bilateral examination),
  * Intraocular pressure (bilateral examination)
  * Measurement of systolic and diastolic blood pressure
  * Heart rate measurement Exercise testing will be performed on bicycle measuring session with 10 minutes at moderate intensity ( 30% OF MPA), 10 minutes at sustained intensity ( 50% of MPA) and 3 minutes at maximum (70% of MPA).
  The theoretical maximal aerobic power was calculated by a mathematical formula.
Other: Examination of pressures after stopping the exercise — In healthy patients performing aerobic physical exercise in the Department of Sports Medicine, the investigators will perform different examinations :
  * Macular and peri-papillary OCT in EDI mode (bilateral examination),
  * Intraocular pressure (bilateral examination)
  * Measurement of systolic and diastolic blood pressure
  * Heart rate measurement Exercise testing will be performed on bicycle measuring session with 10 minutes at moderate intensity ( 30% OF MPA), 10 minutes at sustained intensity ( 50% of MPA) and 3 minutes at maximum (70% of MPA).
  The theoretical maximal aerobic power was calculated by a mathematical formula.

SUMMARY:
Study the change of retrofoveolar choroidal thickness measured by optical coherence tomography during aerobic exercise inducing an increase in systolic blood pressure in healthy subjects.Ten healthy participants will perform an exercise (riding a bicycle ergometer) and will be examined with EDI-OCT. Each participant will be scanned before exercise, during the exercise and afterwards at 0 and 5 min. Each OCT measurement will be coupled to the arterial blood pressure evaluation.

DETAILED DESCRIPTION:
Currently there is a growing interest in the study of the choroid in the pathogenesis of many ocular pathologies such as central serous chorioretinitis1, age-related macular degeneration, diabetic retinopathy, and myopia. Moreover, the recent development of new imaging methods allows the exploration of the normal and pathological processes of the choroid. In particular, the Enhanced Depth Imaging (EDI) mode in Optical Coherence Tomography (OCT) provides cross-sectional imaging of the choroid and in vivo measurement of its thickness. Understanding the factors that would modify the choroidal thickness would make it possible to better understand the pathophysiology of many chorioretinal pathologies and would help to guide therapeutics in the future.

However, systemic changes induced by physical activity, and in particular changes in systolic blood pressure, could be responsible for changes in the choroidal blood flow and thus in the choroidal thickness. The study consists in testing ten patients who will perform an exercise testing as part of the practice of a sportive activity. Patients will undergo an OCT in EDI mode to measure the retrofoveolar choroidal thickness during the exercise.

Each OCT image will be coupled to the evaluation of blood pression and heart rate.

Patients are treated in the usual way but the study is an interventional study, with minimal risks and constraints, because of the imaging (OCT image in EDI mode).

ELIGIBILITY:
Inclusion Criteria:

* Male patients wishing to perform a standardized aerobic exercise stress test Best - Corrected visual acuity ≥ 10/10 (Monoyer scale)
* Absence of ocular pathologies
* Absence of previous ocular surgery
* Refraction between -4 diopters and +4 diopters
* Absence of alcohol or drug abuse
* Absence of systemic pathologies
* Absence of regular doping ;

Exclusion Criteria :

* History of ocular pathologies, intraocular surgery
* Macular or papillary abnormality seen at OCT
* History of systemic pathology such as high blood pressure, diabetes
* Exercise <72 hours
* Intake of coffee or tea <48 hours
* High myopia (axial length> 26mm) or high hyperopia (axial length <19mm) -
* Professional athlete ;Sedentary patient doing sports less than twice a month ; smocking <24 hours
* Pharmacological pupillary dilation <72 hours

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Measurement of macular choroidal thickness before, during and after standardized aerobic exercise inducing a standardized increase in arterial systolic pressure | 1 day
  Measurement of macular choroidal thickness before, during and after standardized aerobic exercise inducing a standardized increase in arterial systolic pressure: the choroidal thickness will be determined thanks to the OCT as the vertical distance between the outer line of the pigmentary epithelium and the internal line of the sclera centered on the fovea thanks to the EDI measurement mode.

SECONDARY OUTCOMES:
Measurement of systolic and diastolic blood pressure | 2 hours (during the consultation)
  Before, during and after the effort The effort is with sustained intensity and maximum intensity. It's a standardized aerobic exercise inducing an increase in systolic arterial blood pressure and arterial diastolic blood pressure.
  An OCT examination in EDI mode focused on the systolic and diastolic blood pressure are taken before the start of the exercise test, during the phase of moderate effort, sustained and maximum, at the end of the effort and 5 minutes after stopping.
Measurement of intraocular pressure | 2 hours (during the consultation)
  Measurement of intraocular pressure systolic and diastolic : Before, during and after the effort The effort with sustained intensity and maximum intensity. It's a standardized aerobic exercise inducing an increase in systolic arterial blood pressure and arterial diastolic blood pressure.
  An OCT examination in EDI mode focused on the macular and peripapillary region the systolic and diastolic blood pressure are taken before the start of the exercise test, during the phase of moderate effort, sustained and maximum, at the end of the effort and 5 minutes after stopping.
Analysis of the peripapillary choroid in OCT | 2 hours (during the consultation)
  Before, during and after the effort Patients presenting for consultation to perform an exercise test in the sports medicine department benefit from an ophthalmological consultation with measurement : The effort with sustained intensity and maximum intensity. It's a standardized aerobic exercise inducing an increase in systolic arterial blood pressure and arterial diastolic blood pressure.
  An OCT examination in EDI mode focused on the macular and peripapillary region during the phase of moderate effort, sustained and maximum, at the end of the effort and 5 minutes after stopping.
Analysis of the retinal vascular caliber on the infrared image of the OCT | 2 hours (during the consultation)
  Analysis of the retinal vascular caliber on the infrared image of the OCT : Before, during and after the effort The effort with sustained intensity and maximum intensity. It's a standardized aerobic exercise inducing an increase in systolic arterial blood pressure and arterial diastolic blood pressure.
  An OCT examination in EDI mode focused on the macular and peripapillary region during the phase of moderate effort, sustained and maximum, at the end of the effort and 5 minutes after stopping.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent SOLER, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No